CLINICAL TRIAL: NCT06044194
Title: Evaluation of the Effect of Liposomal L-Arg and Vit C Integration on Mitochondrial Function in Patients With Heart Failure
Acronym: Mito-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: DAMOR Farmaceutici S.p.a. (Unknown)
Responsible Party: Principal Investigator, Stefano Carugo, Director of the Department of Cardio-Thoracic-Vascular Diseases, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3189
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Mitochondrial; PBMC; L-Arg; Vit C
MeSH Terms: conditions — Heart Failure | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: Pilot, monocentric, national, non-pharmacological, prospective, double-blind randomized trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Placebo Comparator): Once the diagnosis of heart failure is established, patients will be randomized into a double-blind treatment to receive with a 1:1 ratio an oral supplement of 1.66 g L-arginine and 500 mg of liposomal vitamin C once a day (Bioarginine. C , Pharmaceutical Damor) for 3 months (treatment group)
  Interventions: Drug: L-arginine and liposomal vitamin C
- Control group (No Intervention): Once the diagnosis of heart failure is established, patients will be randomized into a double-blind treatment to receive with a 1:1 ratio an oral supplement of Placebo for 3 months (control group)

INTERVENTIONS:
Drug: L-arginine and liposomal vitamin C — Once the diagnosis of heart failure is established, patients will be randomized into a double-blind treatment to receive with a 1:1 ratio an oral supplement of 1.66 g L-arginine and 500 mg of liposomal vitamin C once a day (Bioarginine. C , Pharmaceutical Damor) for 3 months (treatment group) or an oral supplement of Placebo once a day for 3 months (control group)
  Arms: Treatment group

SUMMARY:
Pilot study to assess the effect of L-Arg and Vit C liposomal supplementation on mitochondrial function in patients with heart failure, through analysis of the viability of mitochondria isolated from peripheral blood of mononucleate cells (PBMC).

DETAILED DESCRIPTION:
Pilot, monocentric, national, non-pharmacological, prospective, double-blind randomized trial.

The primary objective of this study is to assess the effect of liposomal L-Arg and Vit C supplementation on mitochondrial function in patients with heart failure, by analysis of the viability of mitochondria isolated from peripheral blood of mononucleate cells (PBMC). Mitochondrial respiratory function of PBMC (in extensive lymphocytes and monocytes) is readily available. These cells are involved in many inflammatory diseases, including those driven by episodes of ischemia-reperfusion, which play a key role in cardiovascular alterations. In particular, the recruitment of T cells and myocardial infiltration are well described during ischemic and non-sischemic heart failure, so the mitochondrial function of PBMC could play a significant role in this immune disorderrelated during heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of heart failure with preserved EF 45%.

Exclusion Criteria:

* Age <18 years
* Left ventricular ejection fraction <45%
* Valvular heart disease
* Previous myocardial infarction or coronary heart disease
* Hypertension
* Diabetes mellitus
* Intolerance to L-arginine and liposomal vitamin C
* Pregnancy
* Lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of liposomal L-Arg and Vit C | 3 months
  The primary objective of this study is to assess the effect of liposomal L-Arg and Vit C supplementation on mitochondrial function in patients with heart failure, by analysis of the viability of mitochondria isolated from peripheral blood of mononucleate cells (PBMC).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No